CLINICAL TRIAL: NCT02074267
Title: Clinical Study for Assessment of the Efficacy of Gabapentin (Carbatin and Neurontin) in Patients With Neuropathy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nang Kuang Pharmaceutical Co., Ltd. (Industry)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S08174
Record Dates: First submitted 2014-02-24; First posted 2014-02-28 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2020-07

CONDITIONS: Neuropathy; Pain
MeSH Terms: conditions — Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Carbatin (Experimental): Carbatin is initiated at 100 mg at night and slowly titrated to 300~800 mg three times/day over 4 to 25 days
  Interventions: Drug: Carbatin
- Neurontin (Active Comparator): Neurontin is initiated at 100 mg at night and slowly titrated to 300~800 mg three times/day over 4 to 25 days
  Interventions: Drug: Neurontin

INTERVENTIONS:
Drug: Carbatin — Carbatin® or Neurontin® is initiated at 100 mg at night and slowly titrated to 300~800 mg three times/day over 4 to 25 days.
  The dose of Carbatin® or Neurontin® taken by each patient will amount to 100 to 2400 mg /day oral if the pain intensity reaches a VAS score ≧4. The maintenance dose of Carbatin® or Neurontin® will throughout for at least 14 days of the treatment period.
  Arms: Carbatin
Drug: Neurontin — Carbatin® or Neurontin® is initiated at 100 mg at night and slowly titrated to 300~800 mg three times/day over 4 to 25 days.
  The dose of Carbatin® or Neurontin® taken by each patient will amount to 100 to 2400 mg /day oral if the pain intensity reaches a VAS score ≧4. The maintenance dose of Carbatin® or Neurontin® will throughout for at least 14 days of the treatment period.
  Arms: Neurontin

SUMMARY:
The purpose of this study is to assess the efficacy of Gabapentin (Carbatin & Neurontin) in patients with neuropathy pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been diagnosed the disease of neuropathy pain arising from diabetic peripheral neuropathy, postherpetic neuralgia, traumatic/surgical nerve injury, incomplete spinal cord injury, or trigeminal neuralgia and if they have a mean weekly pain score of at least 4 on the 100-mm visual analog scale (VAS) of the Short-Form McGill Pain Questionnaire (SF-MPQ) completed a screening / baseline period before randomization. Additional disease-specific inclusion criteria are listed in Table 1.
* Subjects must be 20 years of age or older.

Exclusion Criteria:

* Subjects who are pregnant, lactating or of childbearing potential not using effective contraceptives.
* Subjects who have a clinically significant or unstable medical or psychiatric condition.
* Subjects who are known of hypersensitivity to Gabapentin.
* Serum creatinine > 1.5 times the upper limit of normal
* Subjects who have received nerve blocks or acupuncture for pain relief within four weeks before a screening / baseline period.
* Subjects who have the presence of chronic pain other than the target pain being studied (unless the chronic pain is in a different body region than the target pain and its intensity is not greater than that of the target pain).
* Subjects who have received nondrug therapies or any special procedures for the relief of the target pain within two weeks before a baseline visit.
* Subjects who are using the following agents within 30 days prior to screening: antidepressants, opioids, other anticonvulsants, local anaesthetic injections or any investigational drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain intensity using the visual analog scale (VAS) | up to six weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nang Kuang Pharmaceutical Co., LTD, Tainan, Taiwan